CLINICAL TRIAL: NCT04191083
Title: Assessment of the Effects of Motor Imagery and Action Observation on Motor Learning in Healthy Subjects: a Randomized Controlled Trial
Brief Title: Motor Imagery and Action Observation on Motor Learning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: uammadrid20
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Motor Learning
Keywords: Motor imagery; Action observation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Motor Imagery (Experimental)
  Interventions: Behavioral: Motor imagery
- Double Time Motor Imagery (Experimental)
  Interventions: Behavioral: Double time motor imagery
- Action observation (Experimental)
  Interventions: Behavioral: Action observation
- Placebo group (Placebo Comparator)
  Interventions: Behavioral: Placebo intervention

INTERVENTIONS:
Behavioral: Motor imagery — This group will perform motor imagery training on motor learning of different motor tasks
  Arms: Motor Imagery
Behavioral: Double time motor imagery — This group will perform motor imagery training by doubling the intervention time to the motor imagery group on motor learning of various motor tasks.
  Arms: Double Time Motor Imagery
Behavioral: Action observation — This group will perform action observation training on motor learning of various motor tasks.
  Arms: Action observation
Behavioral: Placebo intervention — This group will watch a video of a landscape without the presence of people.
  Arms: Placebo group

SUMMARY:
This study evaluates the influence of motor imagery and action observation on motor learning

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic subjects
* men and women between 18 and 65 years of age
* participants with no systemic, neurological, cognitive or psychological disease.

Exclusion Criteria:

* underage participants
* presence of systemic pathology, pain and/or weakness that prevents the protocol
* participants who have undergone an operation in the spine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
The Purdue Pegboard test | Change from hit ratio in a manual skill between baseline and 1 week
  This main variable will be composed by the learning of a sequence of digital movements

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No